CLINICAL TRIAL: NCT00664079
Title: Thyroid Hormone Deficiency in Critically Ill Children
Brief Title: Thyroid Hormones in Critically Ill Children
Acronym: Thyroid
Status: Terminated | Type: Observational
Why Stopped: Sluggish enrollment.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-10-4547
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2008-07

CONDITIONS: Hypotension; Respiratory Failure
Keywords: Thyroid Deficiency; Thyroid Stimulating Hormone
MeSH Terms: conditions — Hypotension; Respiratory Insufficiency; Hypothyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who are receiving vasoactive medications and/or are mechanically ventilated.
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — 17 mls of blood will be drawn over a 5 day period from either a central venous catheter/arterial line or with scheduled phlebotomy. The following labs will be run tT3, fT3, rT#, tT4, fT4, TSH, and tyrosine.
  Other Names: Critically Ill Children; Vasoactive Infusions in Children; Mechanical Venilation in Children; Thyroid Deficiency

SUMMARY:
Thyroid hormones are substances naturally made by the body and are important to many of your body's basic functions such as breathing and brain function. We are investigating whether or not these hormones are at lower levels in critically ill children which could lead to further health problems. We hope to get a better understanding of hormone levels and their effects on critically ill children to better help other children in the future.

DETAILED DESCRIPTION:
We hypothesize that critically ill children that require vasoactive infusions and/or invasive mechanical ventilation have thyroid hormone alterations. We will measure TSH, tT3, fT3, rT3, tT4, fT4, adn tyrosine concentrations in critically ill children with hypotension and/or respiratory failure and correlate thyroid hormone alterations to severity of illness, intensity of therapeutic interventions, and associated morbidity and mortality by using clinical outcomes parameters.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Age of less than 12 months and less than or equal to 18
* Patient must weigh greater than 10 kgs.
* Patients must require vasoactive infusions and/or mechanical ventilation.
* Patients must be enrolled within 24 hours of meeting eligibility.

Exclusion Criteria:

* Patient with known or presumed pre-existing thyroid disease will be excluded
* Patients who receive thyroid supplementation will be excluded
* Patients with known or presumed hypothalamic and/or pituitary dysfunction that have thyroid hormone concentration abnormalities not related to an acute illness.
* Patients who are intubated for airway protection only.
* Patients intubated for neuromuscular disease
* Pregnant patients.
* Patients receiving amiodarone supplementation
* Patients who received blood product transfusions equaling more than 1/2 of their blood volume.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are admitted to the Pediatric Intensive Care Unit at the Children's Hospital of Philadelphia will be approached if they meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Certain critically ill children requiring vasoactive infusions and/or mechanical ventilation have low concentrations of tT3, fT3, tT4, fT4, elevated rT3, adn inappropriate low/normal TSH. | When patient has completed the study.

SECONDARY OUTCOMES:
Critically ill children with more severe thyroid hormone deficiencies will have greater severity of illness, intensity of therapeutic intervention, organ dysfunction, and increased morbidity and mortality. | When study is completed.
Critically ill children requiring vasoactive infusions and/or mechanical ventilation are a population in the ICU that has thyroid hormone pertubation and significant morbidity and mortality. | At completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States